CLINICAL TRIAL: NCT02688088
Title: Effects of Multiple Doses of Abemaciclib on the Pharmacokinetics of Cytochrome P450 (CYP) 1A2, CYP2C9, CYP2D6, and CYP3A Substrates (Caffeine, Warfarin, Dextromethorphan, and Midazolam) in Cancer Patients
Brief Title: A Study of Abemaciclib in Participants With Cancer That is Advanced or Has Spread to Another Part(s) of the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15537; I3Y-MC-JPCB (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-04-01

CONDITIONS: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Caffeine; Warfarin; Dextromethorphan; Midazolam; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Drug Cocktail - Period 1 (Active Comparator): Single dose of drug cocktail: 100 milligram (mg) caffeine,10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 1 in Period 1.
  Interventions: Drug: Drug Cocktail
- 200 mg Abemaciclib + Drug Cocktail - Period 2 (Experimental): 200 mg Abemaciclib administered orally every 12 hours (Q12H) on Days 1 - 12 in Period 2 with a single dose of drug cocktail: 100 mgcaffeine,10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 8 in Period 2.
  Interventions: Drug: Drug Cocktail; Drug: Abemaciclib
- 200 mg Abemaciclib - Period 3 (Experimental): 200 mg Abemaciclib administered orally Q12H on Days 13 to 28 in Period 3. Participants may continue to receive abemaciclib until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib
- 200 mg Abemaciclib - Period 4 (Experimental): 200 mg Abemaciclib administered orally Q12H on Days 1 to 28 in Period 4. Participants may continue to receive abemaciclib until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib
- Safety Extension Period (Experimental): 200 mg Abemaciclib administered orally Q12H on Days 1 to 28 onwards in extension period. Participants may continue to receive abemaciclib until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Drug Cocktail — Administered orally
  Other Names: Caffeine + Warfarin + Dextromethorphan + Midazolam
  Arms: 200 mg Abemaciclib + Drug Cocktail - Period 2; Drug Cocktail - Period 1
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: 200 mg Abemaciclib + Drug Cocktail - Period 2; 200 mg Abemaciclib - Period 3; 200 mg Abemaciclib - Period 4; Safety Extension Period

SUMMARY:
This study is known as a "drug interaction study" and is being done to see how abemaciclib may affect the blood levels of a drug mixture of commonly used drugs (caffeine, warfarin, dextromethorphan, and midazolam) when taken in combination with abemaciclib. Each participant will complete screening and four study periods in a fixed sequence, with the option to continue to receive abemaciclib in a safety extension phase. All participants will complete a safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic
* Have adequate organ function
* Have a performance status of ≤2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous therapies for cancer (including chemotherapy, radiotherapy, immunotherapy, cancer-related hormone therapy, and investigational therapy) for at least 21 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents prior to receiving study drug and have recovered from the acute effects of therapy(treatment related toxicity resolved to baseline), except for residual alopecia

Exclusion Criteria:

* Require treatment with inducers or inhibitors of cytochrome P450 (CYP)1A2, CYP2C9, CYP2D6, and CYP3A within 14 days before the first dose of study drug through the end of Period 2
* History or presence of significant bleeding disorders
* Have known active uncontrolled or symptomatic CNS metastases
* Have a primary liver tumor
* Have lymphoma or leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2018-02-04 (Actual); Study Completion 2021-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - IU Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Hospital, Fairway, Kansas
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - South Texas Accelerated Research Therapeutics, LCC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of Abemaciclib in Participants With Cancer That is Advanced or Has Spread to Another Part(s) of the Body — https://trials.lillytrialguide.com/en-US/trial/6XBlVQ9rvUSAoYsMwsICsu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Abemaciclib dose adjustments were allowed due to drug-related toxicity. Before the start of each cycle, drug-related toxicities must have resolved to either baseline or at least Grade 2. Participants not recovered from toxicities within 14 days were discontinued from the study. For Period 2, if abemaciclib dose adjustments occurred, dosing with the drug cocktail was permitted to be delayed to allow for adequate exposure.
Groups:
- Drug Cocktail - Period 1: Single dose of drug cocktail: 100 mg caffeine, 10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 1 in Period 1.
- 200 mg Abemaciclib + Drug Cocktail - Period 2: 200 mg Abemaciclib administered orally every 12 hours (Q12H) on Days 1 to 12 in Period 2.
  Single dose of drug cocktail: 100 mg caffeine, 10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 8 in Period 2.
- 200 mg Abemaciclib - Period 3: 200 mg Abemaciclib administered orally Q12H on Days 13 to 28 in Period 3.
  .
- 200 mg Abemaciclib Period - 4: 200 mg Abemaciclib administered orally Q12H on Days 1 to 28 in Period 4.
- Abemaciclib Safety Extension Period: 200 mg Abemaciclib administered orally Q12H on Days 1 to 28 onwards in extension period.
Period: Single Dose Drug Cocktail - Period 1
Arm/Group | Drug Cocktail - Period 1 | 200 mg Abemaciclib + Drug Cocktail - Period 2 | 200 mg Abemaciclib - Period 3 | 200 mg Abemaciclib Period - 4 | Abemaciclib Safety Extension Period
Started | 44 | 0 | 0 | 0 | 0
Received One Dose of Drug Cocktail | 44 | 0 | 0 | 0 | 0
Completed | 44 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Abemaciclib + Drug Cocktail - Period 2
Arm/Group | Drug Cocktail - Period 1 | 200 mg Abemaciclib + Drug Cocktail - Period 2 | 200 mg Abemaciclib - Period 3 | 200 mg Abemaciclib Period - 4 | Abemaciclib Safety Extension Period
Started | 0 (Participants received Drug Cocktail in Period 1 only.) | 44 (Participants entered Period 2 to receive Abemaciclib on Days 1 to 12 and Drug Cocktail on Day 8.) | 0 | 0 | 0
Received at Least One Dose of Study Drug | 0 | 42 | 0 | 0 | 0
Completed | 0 | 37 | 0 | 0 | 0
Not Completed | 0 | 7 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0
Period: Abemaciclib Days 13 to 28 - Period 3
Arm/Group | Drug Cocktail - Period 1 | 200 mg Abemaciclib + Drug Cocktail - Period 2 | 200 mg Abemaciclib - Period 3 | 200 mg Abemaciclib Period - 4 | Abemaciclib Safety Extension Period
Started | 0 | 0 (Participants completed Period 2.) | 37 (Participants continue Abemaciclib in Period 3.) | 0 | 0
Received at Least One Dose of Study Drug | 0 | 0 | 36 | 0 | 0
Completed | 0 | 0 | 29 | 0 | 0
Not Completed | 0 | 0 | 8 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 7 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Period: Abemaciclib Days 1 to 28 - Period 4
Arm/Group | Drug Cocktail - Period 1 | 200 mg Abemaciclib + Drug Cocktail - Period 2 | 200 mg Abemaciclib - Period 3 | 200 mg Abemaciclib Period - 4 | Abemaciclib Safety Extension Period
Started | 0 | 0 | 0 (Participants completed Abemaciclib Period 3.) | 29 (Participants continued to receive Abemaciclib in Period 4.) | 0
Completed | 0 | 0 | 0 | 21 | 0
Not Completed | 0 | 0 | 0 | 8 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 7 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Period: Abemaciclib Safety Extension Period
Arm/Group | Drug Cocktail - Period 1 | 200 mg Abemaciclib + Drug Cocktail - Period 2 | 200 mg Abemaciclib - Period 3 | 200 mg Abemaciclib Period - 4 | Abemaciclib Safety Extension Period
Started | 0 | 0 | 0 | 0 (Participants completed Period 4.) | 18 (Participants had option of continuing Abemaciclib in Safety Extension Period.)
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 0 | 18
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 18
Not completed — Met Discontinuation Criteria | 0 | 0 | 0 | 0 | 18

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of drug cocktail.
Groups:
- Overall: A single dose of drug cocktail was administered on Day 1 of Period 1. Abemaciclib 200 mg was administered Q12H starting on Day 1 of Period 2 with coadministration of drug cocktail on Day 8. Participants continued to receive 200 mg abemaciclib (or modified dose as required) Q12H up to 16 days in Period 3 and up to 28 days in Period 4. Participants could participate in a safety extension phase in which they received 200 mg abemaciclib (or modified dose as required) Q12H until discontinuation criteria are met.
Arm/Group | Overall
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 40
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Caffeine
Description: Maximum concentration of caffeine after single dose of drug cocktail on Day 1 in Period 1 and in combination with Abemaciclib on Day 8 in Period 2.
Time Frame: Days 1 and 8: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, and 48 hours (hr) Postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 100 mg Caffeine: Single oral dose of 100 mg caffeine administered orally on Day 1 in Period 1.
- Abemaciclib + 100 mg Caffeine: 200 mg Abemaciclib administered orally Q12H on Days 1 to 12 in Period 2.
  Single dose of drug cocktail: 100 mg caffeine, 10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 8.
Arm/Group | 100 mg Caffeine | Abemaciclib + 100 mg Caffeine
Number analyzed (Participants) | 39 | 32
nanograms per milliliter (ng/mL) | 2890 (29) | 2950 (33)
Statistical Analysis 1: Comparison: 100 mg Caffeine vs Abemaciclib + 100 mg Caffeine; Test type: Superiority; Ratio of Geometric LS Means = 1.01, 90% CI 2-sided [0.965 to 1.06]

2. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) S-Warfarin
Description: Maximum concentration of S-warfarin after single dose of drug cocktail on Day 1 in Period 1and in combination with Abemaciclib on Day 8 in Period 2.
Time Frame: Days 1 and 8: Predose, 0.5 1, 2, 3, 4, 6, 8, 12, 48, 72, 96 hr Postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 10 mg Warfarin: 10 mg warfarin administered orally on Day 1 in Period 1.
- 200 mg Abemaciclib + 10 mg Warfarin: 200 mg Abemaciclib administered orally Q12H on Days 1 to 12 in Period 2.
  Single dose of drug cocktail: 100 mg caffeine, 10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 8.
Arm/Group | 10 mg Warfarin | 200 mg Abemaciclib + 10 mg Warfarin
Number analyzed (Participants) | 44 | 30
ng/mL | 561 (35) | 526 (35)
Statistical Analysis 1: Comparison: 10 mg Warfarin vs 200 mg Abemaciclib + 10 mg Warfarin; Test type: Superiority; Ratio of Geometric LS Means = 0.935, 90% CI 2-sided [0.871 to 1.00]

3. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Dextromethorphan
Description: Maximum concentration of dextromethorphan after single dose of drug cocktail on Day 1 of Period 1 and in combination with Abemaciclib on Day 8 in Period 2.
Time Frame: Days 1 and 8: Predose, 1, 2, 4, 6, 8, 10, 24, 48, 72 hr postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 30 mg Dextromethorphan: 30 mg dextromethorphan administered orally on Day 1 in Period 1.
- 200 Abemaciclib + 30 mg Dextromethorphan: 200 mg Abemaciclib administered orally Q12H on Days 1 to 12 in Period 2.
  Single dose of drug cocktail: 100 mg caffeine, 10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 8 in Period 2.
Arm/Group | 30 mg Dextromethorphan | 200 Abemaciclib + 30 mg Dextromethorphan
Number analyzed (Participants) | 43 | 36
ng/mL | 3.18 (182) | 3.30 (164)
Statistical Analysis 1: Comparison: 30 mg Dextromethorphan vs 200 Abemaciclib + 30 mg Dextromethorphan; Test type: Superiority; Ratio of Geometric LS Means = 1.05, 90% CI 2-sided [0.898 to 1.22]

4. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Midazolam
Description: Maximum concentration of midazolam after single dose of drug cocktail on Day 1 of Period 1 and in combination with Abemaciclib on Day 8 in Period 2.
Time Frame: Days 1 and 8: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hr Postdose
Population: All subjects who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 0.2 mg Midazolam (Drug Cocktail): Single dose of 0.2 mg midazolam administered orally on Day 1 in Period 1.
- 200 mg Abemaciclib + 0.2 mg Midazolam: 200 mg Abemaciclib administered orally Q12H on Days 1 to 12 in Period 2.
  Single dose of drug cocktail: 100 mg caffeine, 10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 8 in Period 2.
Arm/Group | 0.2 mg Midazolam (Drug Cocktail) | 200 mg Abemaciclib + 0.2 mg Midazolam
Number analyzed (Participants) | 44 | 39
ng/mL | 2.12 (54) | 1.75 (48)
Statistical Analysis 1: Comparison: 0.2 mg Midazolam (Drug Cocktail) vs 200 mg Abemaciclib + 0.2 mg Midazolam; Test type: Superiority; Ratio of Geometric LS Means = 0.845, 90% CI 2-sided [0.760 to 0.940]

5. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve [AUC(0-infinity)] of Caffeine
Description: PK: AUC zero to infinity of caffeine after single dose of drug cocktail on Day 1 in Period 1 and in combination with Abemaciclib on Day 8 in Period 2.
Time Frame: Days 1 and 8: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 hr Postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Groups:
- 100 mg Caffeine: Single dose of 100 mg caffeine administered orally on Day of Period 1.
- 200 mg Abemaciclib + 100 mg Caffeine: 200 mg Abemaciclib administered orally Q12H on Days 1 to 12 in Period 2.
  Single dose of drug cocktail: 100 mg caffeine, 10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 8.
Arm/Group | 100 mg Caffeine | 200 mg Abemaciclib + 100 mg Caffeine
Number analyzed (Participants) | 37 | 30
nanograms*hour per milliliter (ng*h/mL) | 32500 (72) | 47100 (89)
Statistical Analysis 1: Comparison: 100 mg Caffeine vs 200 mg Abemaciclib + 100 mg Caffeine; Test type: Superiority; Ratio of Geometric LS Means = 1.56, 90% CI 2-sided [1.35 to 1.81]

6. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve [AUC(0-infinity)] of S-Warfarin
Description: AUC (zero to infinity) of S-warfarin after single dose of drug cocktail on Day 1 in Period 1 and in combination with Abemaciclib on Day 8 in Period 2.
Time Frame: Days 1 and 8: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hr Postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- 10 mg Warfarin: Single dose 10 mg warfarin administered orally on Day of Period 1.
Arm/Group | 10 mg Warfarin | 200 mg Abemaciclib + 10 mg Warfarin
Number analyzed (Participants) | 44 | 30
ng*h/mL | 21400 (43) | 20600 (40)
Statistical Analysis 1: Comparison: 10 mg Warfarin vs 200 mg Abemaciclib + 10 mg Warfarin; Test type: Superiority; Ratio of Geometric LS Means = 1.04, 90% CI 2-sided [0.956 to 1.13]

7. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve [AUC(0-infinity)] of Dextromethorphan
Description: PK: AUC (zero to infinity) of dextromethorphan after single dose of drug cocktail on Day 1 in Period 1 and in combination with Abemaciclib on Day 8 in Period 2.
Time Frame: Days 1 and 8: 1, 2, 4, 6, 8, 10, 24, 48, 72 hr Postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- 30 mg Dextromethorphan: Single dose 30 mg administered orally on Day 1 of Period 1.
- 200 mg Abemaciclib + 30 mg Dextromethorphan: 200 mg Abemaciclib administered orally Q12H on Days 1 to 12 in Period 2.
  Single dose of drug cocktail: 100 mg caffeine, 10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 8.
Arm/Group | 30 mg Dextromethorphan | 200 mg Abemaciclib + 30 mg Dextromethorphan
Number analyzed (Participants) | 42 | 35
ng*h/mL | 32.6 (316) | 32.1 (238)
Statistical Analysis 1: Comparison: 30 mg Dextromethorphan vs 200 mg Abemaciclib + 30 mg Dextromethorphan; Test type: Superiority; Mean Difference (Final Values) = 0.976, 90% CI 2-sided [0.805 to 1.18]

8. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve [AUC(0-infinity)] of Midazolam
Description: PK: AUC (zero to infinity) of midazolam after single dose of drug cocktail on Day 1 in Period 1 and in combination with Abemaciclib on Day 8 in Period 2.
Time Frame: Days 1 and 8: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hr Postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- 0.2 mg Midazolam: Single dose 0.2 mg midazolam administered orally on Day 1 of Period 1.
- 200 mg Abemaciclib + 0.2 mg Midazolam: 200 mg Abemaciclib administered orally Q12H on Days 1 to 12 in Period 2.
  Single dose of drug cocktail: 100 mg caffeine, 10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 8.
Arm/Group | 0.2 mg Midazolam | 200 mg Abemaciclib + 0.2 mg Midazolam
Number analyzed (Participants) | 44 | 37
ng*h/mL | 7.34 (74) | 6.03 (63)
Statistical Analysis 1: Comparison: 0.2 mg Midazolam vs 200 mg Abemaciclib + 0.2 mg Midazolam; Test type: Superiority; Ratio of Geometric LS Means = 0.867, 90% CI 2-sided [0.775 to 0.972]

9. Secondary Outcome: Mean Change From Baseline at 24 Hours in Systolic and Diastolic Blood Pressure in Period 1
Description: Mean change from predose in systolic and diastolic blood pressure (BP) over 24 hours (h) postdose following single dose drug cocktail in Period 1.
Time Frame: Day 8: Baseline, 24 h postdose
Population: All subjects who received at least one dose of study drug and had at least one postdose safety assessment.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Groups:
- Drug Cocktail Period 1: Single dose of drug cocktail: 100 mg caffeine, 10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 1 in Period 1.
Arm/Group | Drug Cocktail Period 1
Number analyzed (Participants) | 44
millimeter of mercury (mmHg)
  Systolic BP | -2.5 (13.9)
  Diastolic BP | -0.7 (10.1)

10. Secondary Outcome: Mean Change From Baseline at 24 Hours in Pulse Rate in Period 1
Description: Mean change from baseline in pulse rate over 24 hours (h) postdose following single dose drug cocktail in Period 1.
Time Frame: Day 8: Baseline, 24 h postdose
Population: All subjects who received at least one dose of study drug and had at least one postdose safety assessment.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Drug Cocktail Period 1
Number analyzed (Participants) | 44
Beats per minute (bpm) | -1.3 (11.1)

11. Secondary Outcome: Mean Change From Baseline at 24 Hours in Systolic and Diastolic Blood Pressure in Period 2
Description: Mean change from baseline in systolic and diastolic blood pressure (BP) over 24 hours (h) postdose following single dose of abemaciclib in Period 2, Day 1.
Time Frame: Day 1: Baseline, 24 h postdose
Population: All subjects who received at least one dose of study drug and had at least one postdose safety assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- 200 mg Abemaciclib: 200 mg Abemaciclib administered orally Q12H on Days 1 to 12 in Period 2.
Arm/Group | 200 mg Abemaciclib
Number analyzed (Participants) | 41
mmHg
  Systolic BP | -7.8 (15.2)
  Diastolic BP | -1.8 (10.4)

12. Secondary Outcome: Mean Change From Baseline at 24 Hours in Pulse Rate in Period 2
Description: Mean change from baseline in pulse rate over 24 hours (h) postdose following single dose drug cocktail in Period 2, Day 1.
Time Frame: Day 1: Baseline, 24 h postdose
Population: All subjects who received at least one dose of study drug and had at least one postdose safety assessment.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | 200 mg Abemaciclib
Number analyzed (Participants) | 41
bpm | -0.2 (12.5)

13. Secondary Outcome: Mean Change From Baseline at 24 Hours in Systolic and Diastolic Blood Pressure in Period 2
Description: Mean change from baseline in systolic and diastolic blood pressure (BP) at 24 h postdose following 200 mg abemaciclib and drug cocktail.
Time Frame: Day 8: Baseline, 24 h postdose
Population: All subjects who received at least one dose of study drug and had at least one postdose safety assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- 200 mg Abemaciclib + Drug Cocktail: 200 mg Abemaciclib administered orally Q12H on Days 1 to 12 in Period 2.
  Single dose of drug cocktail: 100 mg caffeine, 10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 8.
Arm/Group | 200 mg Abemaciclib + Drug Cocktail
Number analyzed (Participants) | 39
mmHg
  Systolic BP | -11.6 (16.8)
  Diastolic BP | -6.1 (10.5)

14. Secondary Outcome: Mean Change From Baseline at 24 Hours in Pulse Rate in Period 2
Description: Mean change from baseline in pulse rate at 24 h postdose following 200 mg abemaciclib and drug cocktail.
Time Frame: Day 8: Baseline, 24 h postdose
Population: All subjects who received at least one dose of study drug and had at least one postdose safety assessment.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | 200 mg Abemaciclib + Drug Cocktail
Number analyzed (Participants) | 39
bpm | 4.1 (14.9)

ADVERSE EVENTS:
Time Frame: Baseline up to 46 days
Description: All participants who received at least one dose of study drug and have at least one postdose safety assessment.
  As dose adjustments due to toxicity were allowed in Periods 2, 3, and 4, a participant may have entered Period 3 or 4 on a dose level other than 200 mg Abemaciclib. As a result, the number of participants for Periods 3 and 4 differ between the Participant Flow and the Adverse Events section.
Groups:
- 200 mg Abemaciclib - Period 2: 200 mg Abemaciclib administered orally every 12 hours (Q12H) on Days 1 to 12 in Period 2.
- 200 mg Abemaciclib + Drug Cocktail - Period 2: 200 mg Abemaciclib administered orally Q12H on Days 1 to 12 in Period 2. Single dose of drug cocktail: 100 mg caffeine, 10 mg warfarin, 30 mg dextromethorphan, and 0.2 mg midazolam administered orally on Day 8 in Period 2.
- 200 mg Abemaciclib - Periods 3 and 4: 200 mg Abemaciclib administered orally Q12H on Days 13 to 28 in Period 3, and Days 1 to 28 in Period 4.
- Abemaciclib Safety Extension Period: 200 mg Abemaciclib administered orally Q12H until discontinuation criteria are met.
Arm/Group | Drug Cocktail - Period 1 | 200 mg Abemaciclib - Period 2 | 200 mg Abemaciclib + Drug Cocktail - Period 2 | 200 mg Abemaciclib - Periods 3 and 4 | Abemaciclib Safety Extension Period
All-Cause Mortality (participants affected / at risk) | 1/44 | 0/42 | 0/35 | 0/28 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/44 | 3/42 | 2/35 | 6/28 | 2/18
Other Adverse Events (participants affected / at risk) | 22/44 | 33/42 | 26/35 | 25/28 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Cocktail - Period 1 (N=44) | 200 mg Abemaciclib - Period 2 (N=42) | 200 mg Abemaciclib + Drug Cocktail - Period 2 (N=35) | 200 mg Abemaciclib - Periods 3 and 4 (N=28) | Abemaciclib Safety Extension Period (N=18)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Cocktail - Period 1 (N=44) | 200 mg Abemaciclib - Period 2 (N=42) | 200 mg Abemaciclib + Drug Cocktail - Period 2 (N=35) | 200 mg Abemaciclib - Periods 3 and 4 (N=28) | Abemaciclib Safety Extension Period (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 6 (6) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (2) | 2 (2) | 3 (5)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 18 (18) | 11 (11) | 12 (12) | 2 (5)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 8 (9) | 6 (6) | 7 (8) | 4 (5)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 8 (9) | 5 (7) | 7 (9) | 4 (6)
Fatigue (General disorders) | 1 (1) | 6 (6) | 6 (6) | 5 (5) | 3 (3)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oedema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal vein stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 3 (4)
International normalised ratio increased (Investigations) | 7 (7) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 4 (4) | 6 (7) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 4 (5) | 1 (1) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (6) | 0 (0) | 5 (6) | 3 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT02688088/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT02688088/SAP_001.pdf